CLINICAL TRIAL: NCT01013480
Title: An Open Label Extension Study to Evaluate the Safety, Tolerability and Pharmacokinetics of STX209 in Subjects With Fragile X Syndrome
Brief Title: An Open Label Extension Study of STX209 in Subjects With Fragile X Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: all active subjects rolled into 209FX303/NCT01013480
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22002
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2011-03

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — arbaclofen placarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STX209 (Active Comparator)
  Interventions: Drug: Arbaclofen

INTERVENTIONS:
Drug: Arbaclofen — A flexible dose titration will be utilized during the first four weeks to define the optimal titrated dose (OTD) for each subject. Investigators will use clinical judgment to adjust doses to the OTD. The starting dose will be 1 mg BID. The dose may be increased every four to five days to 2 mg BID, 3 mg BID, 5 mg BID and then 10 mg BID
  Other Names: R-baclofen; STX209

SUMMARY:
Study 22001, "A Double-Blind, Placebo-Controlled, Flexible-Dose Evaluation of the Efficacy, Safety, and Tolerability of STX209 in the Treatment of Irritability in Subjects with Fragile X Syndrome" currently is evaluating the efficacy of STX209 (R-baclofen) for management of typical problem behaviors, such as irritability and aggression, in subjects with FXS. This study (22002) will enter subjects who complete Study 22001 into a long-term, open-label study.The open-label extension protocol will provide necessary data on the long-term safety and tolerability of STX209 among subjects with FXS who receive treatment under conditions more closely reflective of their general medical care.

ELIGIBILITY:
Inclusion Criteria:

* Have completed all scheduled visits in protocol 22001 and have shown they can adequately follow the protocol, with sufficient medical justification to continue on open-label treatment with STX209, as assessed by the principal investigator

Exclusion Criteria:

* Subjects with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being.
* The occurrence or continuation of any adverse event or condition during study 22001 that, in the opinion of the Investigator, should exclude the subject from participating in this open-label extension.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Irritability subscale of the Aberrant Behavior Checklist | 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - M.I.N.D. Institute, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - NYS Institute for Basic Research in Developmental Disabilities, Staten Island, New York
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Suburban Research Associates, Media, Pennsylvania
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, PA, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington